CLINICAL TRIAL: NCT02136251
Title: Five Year Outcome Follow-up of Glenoid Anchor Peg Component Fixation Utilizing Autologous Bone Graft in Total Shoulder Arthroplasty.
Brief Title: Total Shoulder Replacement Outcomes With Autologous Bone Graft as Fixator for Glenoid Anchor Peg.
Acronym: Glenoid
Status: Withdrawn | Type: Observational
Why Stopped: Funding was not obtained to complete study
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0067-14-FB
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Arthritis
Keywords: Total Shoulder Arthroplasty; Glenoid anchor peg component fixation; Autologous bone grafting
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- shoulder replacement: Subjects who had shoulder replacement surgery at The University of Nebraska and The Nebraska Medical Center at least 5 or more years ago and autologous bone graft around the anchor-peg glenoid prosthesis was used.

SUMMARY:
We hypothesize that there will be a low incidence of glenoid loosening with a total shoulder arthroplasty using an anchor peg glenoid and autologous bone grafting. In addition, we suggest that the absence of radiolucent lines will correlate with excellent shoulder function.

DETAILED DESCRIPTION:
This will be five year follow-up of glenoid anchor peg component fixation utilizing autologous bone graft in total shoulder arthroplasty. The purpose of this study is to investigate if the use of autologous bone graft around the anchor peg glenoid prosthesis correlates with better shoulder function. Subjects having had this surgery who are five years or more out from surgery will have computed tomography and three plain radiographs to monitor for bony apposition, radiolucent lines and component loosening. These testings are not a study intervention and are for monitoring purposes.

ELIGIBILITY:
Inclusion Criteria:

- Have had a total shoulder replacement with an anchor peg glenoid and autologous bone grafting at the Department of Orthopaedic Surgery at University of Nebraska and The Nebraska Medical Center five years or longer ago.

Exclusion Criteria:

* unable to comprehend the consent form information
* pregnant women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Orthopaedic Surgery clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09 (Estimated); Primary Completion 2015-02-13 (Actual); Study Completion 2015-02-13 (Actual)

PRIMARY OUTCOMES:
Evidence of lower incidence of glenoid loosening and absence of radiolucent lines confirmed by CT and radiographs. | 5 years after surgery
  To investigate if the use of autologous bone graft around the anchor-peg glenoid prosthesis correlates with (1.) bony apposition on computed tomography scans, (2.) decreased radiolucent lines, (3.) a decrease in component loosening, and (4.) better functional outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Teusink, MD, Principal Investigator — University of Nebraska